CLINICAL TRIAL: NCT03980054
Title: A Phase III Study to Evaluate the Efficacy and Safety of Pyrotinib Versus Placebo in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Positive Early or Locally Advanced Breast Cancer After Adjuvant Trastuzumab
Brief Title: A Study of Evaluating The Effects Of Pyrotinib After Adjuvant Trastuzumab In Women With Early Stage Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-BLTN-III-EBC
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Intervention Model Description: Pyrotinib versus Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Pyrotinib (Experimental): Intervention: Drug: Pyrotinib
  Interventions: Drug: Pyrotinib
- Arm Placebo (Placebo Comparator): Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyrotinib — pyrotinib 400 mg, orally once daily for one year
  Arms: Arm Pyrotinib
Drug: Placebo — placebo 400mg, orally once daily for one year
  Arms: Arm Placebo

SUMMARY:
This is a randomised, double-blind multicenter Phase III study for evaluating the efficacy and safety of pyrotinib in women with early stage high-risk breast cancer after adjuvant trastuzumab. The main purpose of this study is to investigate whether pyrotinib can further reduce the risk of recurrence from previously diagnosed HER-2 positive breast cancer after adjuvant treatment with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18 years ≤ age ≤ 75 years；
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive HER2 positive breast cancer.
* Known hormone receptor status.
* Cardiovascular: Baseline left ventricular ejection fraction (LVEF)≥55% measured by Echocardiogram.
* Been treated for early breast cancer with standard of care duration of trastuzumab.
* If been not treated neoadjuvantly, lymph node metastases need to be confirmed by postoperative pathology; if been treated neoadjuvantly , have not reached totally pathologic complete response.
* Signed informed consent form (ICF) .

Exclusion Criteria:

* Positive clinical and radiologic assessments for local or regional recurrence of disease at the time of study entry.
* History of heart disease.
* Bilateral breast cancer.
* Corrected QT (QTc) interval ≥0.47 seconds.
* History of gastrointestinal disease with diarrhea as the major symptom.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1192 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) | From randomization until time of event up to 2 years
  Invasive disease-free survival time is defined as the time from date of randomization until the first invasive disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, distant recurrence and death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | From randomization until time of event up to 2 years
  Disease-free survival time is defined as the time from date of randomization until the first disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, non-breast primary invasive cancer, ductal carcinoma in situ(DCIS),or distant recurrence and death from any cause.
Overall Survival (OS) | up to 2 years
  Overall survival is defined as the time from randomization to death from any cause.
Distance Disease-free Survival (DDFS) | distant recurrence From randomization until time of event up to 2 years
  Distance Disease-free Survival is defined as the time from date of randomization until the first distant recurrence and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Study Chair — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No